CLINICAL TRIAL: NCT01189643
Title: A Pilot Trial of Irinotecan, Temozolomide and Bevacizumab in Combination With Existing High Dose Alkylator Based Chemotherapy for Treatment of Newly Diagnosed Patients With Desmoplastic Small Round Cell Tumor
Brief Title: Irinotecan, Temozolomide and Bevacizumab in Combination With Existing High Dose Alkylator Based Chemotherapy for Treatment of Newly Diagnosed Patients With Desmoplastic Small Round Cell Tumor
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-091
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Sarcoma; Desmoplastic Small Round Cell Tumor (DSRCT)
Keywords: BEVACIZUMAB (AVASTIN); IRINOTECAN (CPT-11) CAMPTOSAR; TEMOZOLOMIDE; DSRCT; 10-091
MeSH Terms: conditions — Sarcoma; Desmoplastic Small Round Cell Tumor | interventions — Irinotecan; Temozolomide; Alkylating Agents

ARMS (1):
- Chemotherapy (Experimental): This is a pilot study to evaluate the acute toxicities and activity of irinotecan, temozolomide, and bevacizumab incorporated into an existing schedule of high dose alkylator based therapy in newly diagnosed patients with DSRCT.
  Interventions: Drug: irinotecan, temozolomide, and bevacizumab incorporated into an existing schedule of high dose alkylator

INTERVENTIONS:
Drug: irinotecan, temozolomide, and bevacizumab incorporated into an existing schedule of high dose alkylator — Two cycles of the investigational combination irinotecan, temozolomide and bevacizumab- will be given followed by conventional chemotherapy with a modified P6 approach and surgical local control. Completion of modified P6 chemotherapy will be followed by a second-look surgery.

SUMMARY:
This study adds irinotecan, temozolomide and bevacizumab to the chemotherapy regimen currently used to treat Desmoplastic small round cell tumor (DSRCT). The investigators are doing this study to find out what effects, good and/or bad, the combination of irinotecan, temozolomide and bevacizumab has on the patient and the DSRCT cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 1 year, less than 30 years
* Newly diagnosed, previously untreated patients with histologically or molecularly confirmed DSRCT
* Adequate hematologic function:
* Absolute neutrophil count ≥ 1,000/mm3
* Platelet count ≥ 100,000/mytm3
* Adequate renal function:
* Normal creatinine for age OR
* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2
* Adequate hepatic function:
* Total bilirubin ≤ 1.5 x the ULN for age
* AST ≤ 2.5 x the ULN for age [in the absence of hepatic involvement of tumor]
* Normal cardiac function
* Shortening fraction greater than or equal to 28% by echocardiogram OR
* Left ventricular ejection fraction (LVEF) greater than or equal to 50% on technetium-99m pertechnetate radionuclide cineangiography (MUGA) or echocardiogram
* Hypertension must be well controlled on stable doses of medication for at least two weeks prior to enrollment.
* Patients must consent to an indwelling central venous catheter.
* Sexually active patients of reproductive potential must be willing to use an effective method of contraception.

Exclusion Criteria:

* Prior chemotherapy or radiotherapy
* Pregnant or breastfeeding females
* Patients with documented chronic non-healing wound, ulcer or bone fracture.
* Incomplete healing from previous oncologic or other major surgery.
* Surgical procedures:

Patients who have undergone major surgery (including open biopsy, thoracotomy, organ resection, exploratory laparotomy, arteriovenous grafts) <28 days prior to enrollment will have bevacizumab dosing delayed as outlined in section 9.1

* Patients must be at least 48 hours from placement of central catheter before receiving first dose of bevacizumab
* Minor surgical procedures (needle/laparoscopic core biopsies) for limited purposes of tissue retrieval will be allowed. Patients should not receive the first planned dose of bevacizumab until the wound is healed and 7 days have elapsed since the procedure.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Thrombosis:
* Patients must not have had a deep venous or arterial thrombosis (non-central venous catheter related) within the last three months prior to study entry.
* Patients with cerebrovascular accident or transient ischemic attack within 6 months of therapy are excluded
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study entry.
* CNS status: Patients must not have known CNS metastases or leptomeningeal disease.

Screening with brain imaging is not required for asymptomatic patients. Proteinuria: Urine protein: creatinine ratio greater than or equal to 1.0

* Uncontrolled hypertension (defined as SBP and/or DBP > 95th percentile for age)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 12 months prior to Day 1
* History of stroke or transient ischemic attack
* Significant vascular (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Known hypersensitivity to any component of bevacizumab

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To define the tolerability | 2 years
  of irinotecan, temozolomide and bevacizumab in patients with newly diagnosed DSRCT
To define adverse event profile | 2 years
  of irinotecan, temozolomide and bevacizumab in patients with newly diagnosed DSRCT

SECONDARY OUTCOMES:
To estimate the response rate of two cycles of irinotecan, temozolomide and bevacizumab | 2 years
  In patients with measurable disease. added to the initial treatment of patients with Desmoplastic small round cell tumor (DSRCT)
To estimate survival | 2 years
  with the addition of irinotecan, temozolomide and bevacizumab to the initial treatment of patients with DSRCT
To estimate time to progression | 2 years
  with the addition of irinotecan, temozolomide and bevacizumab to the initial treatment of patients with DSRCT
To assess use of 18FDG PET-CT | 2 years
  as an early indicator of response in those patients with measurable or evaluable disease

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm